CLINICAL TRIAL: NCT01603732
Title: Evaluation of Maternal B-hemolytic Streptococcal Pharyngeal Exposure in Pregnancies Affected by Congenital Heart Disease(CHD)
Brief Title: Association Between a Mother's Exposure to "Strep Throat" and Her Baby's Developing Heart Disease
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201102410; 5R01HL098634-02 (NIH)
Record Dates: First submitted 2012-05-18; First posted 2012-05-23 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Congenital Heart Disease in Pregnancy
Keywords: Strep exposure and heart defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Confirmation of maternal ß-hemolytic streptococcal & enterovirus infection(s) will be determined from nose and rectal swabs & blood samples assayed for standard marker antibodies to ß-hemolytic streptococcal & enterovirus exposure.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Moms w HLHS or variant: Mom's fetal diagnosis Hypoplastic Left Heart Syndrome/variant
- Moms w/ Other congential heart defect): Moms fetal diagnosis -other congenital heart defects
- Moms-fetal - echo normal: Moms echo fetal diagnosis is normal.
- Random Healthy Moms: Mom with healthy pregnancy.

SUMMARY:
The goal of this study is to find out if there is any association between a mother's exposure to bacteria that normally causes "strep throat" and her baby's developing heart disease/heart defect.

DETAILED DESCRIPTION:
The primary objective of this study is to:

1. measure maternal ß-hemolytic streptococcal carriage as defined by positive throat cultures in the absence of symptoms among Hypoplastic Left Heart Syndrome (HLHS) mothers.
2. define the incidence of positive strep throat cultures among asymptomatic pregnant women, identified at <18 weeks gestation and followed to term.
3. Measure antibodies that may cross react to select valvular/myocardial antigens in HLHS/Congenital Heart Defect(CHD)-other neonates born to mothers in the study
4. determine serum and/or tissue reactivity against antibodies in matched maternal serum.

The secondary objectives of this study is to:

1. measure maternal ß-hemolytic streptococcal serology using standard serology testing among HLHS mothers.
2. determine the history of maternal ß-hemolytic streptococcal exposure using a study questionnaire among HLHS mothers.
3. Determine "baseline" strep serologies and history of strep exposure among a cohort of asymptomatic pregnant women, identified at <18 weeks gestation and followed to term.

   The overall purpose of this study is to evaluate the history of β-hemolytic streptococcal pharyngeal exposure, groups A, G and C ("strep throat") in pregnant women whose pregnancies have been complicated by the diagnosis of congenital heart disease. Our short-term goal is to identify a potential association of an antecedent maternal strep throat exposure in pregnancy to identify a subset of heart defects
4. To determine if co-infections play a role in congenital heart defects

ELIGIBILITY:
Inclusion Criteria:

* For Fetal pts:
* HLHS or variant diagnosis
* Other Congenital Heart Disease
* Greater than or = 20wks gestation
* For Healthy moms:
* No diagnosis of Congenital Heart Disease
* Greater than or = 20wks gestation

Exclusion Criteria:

* For fetal pts & healthy controls:
* Mom less than 18 years old
* Twins or multiple gestations
* Pregnancy affected by 2 or more congenital anomalies( in addition to heart defects)
* Pregnancy affected by OB complications like pre-eclampsia
* Known history of chromosomal anomaly or carrier status
* Pregnancy result of fertility treatment including in vitro fertilization
* Emotionally distress
* Mom received blood transfusion or immunoglobin infusion within 6 months of the pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random Healthy Controls and Moms with fetal care/echos during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Title: Evaluation of Maternal ß-hemolytic Streptococcal Pharyngeal Exposure in Pregnancies Affected by Congenital Heart Disease | 01/15/2010 - 12/31/2014
  History of strep infection using a detailed questionnaire and maternal medical records (primary end-point) and (b) maternal titers of the anti-strep antibody, anti-streptolysin O (ASO) (secondary endpoint).

SECONDARY OUTCOMES:
Title: Evaluation of Maternal ß-hemolytic Streptococcal Pharyngeal Exposure in Pregnancies Affected by Congenital Heart Disease | 01/15/2010 - 12/31/2014
  To determine if mothers of babies with HLHS have a significant history of strep infections

CONTACTS AND LOCATIONS:
Overall Officials: Pirooz Eghtesady, MD,PhD, Principal Investigator — Washington University School of Medicine and St Louis Children's Hospital
Locations (2):
- United States (2):
  - St Louis Childrens Hospital, St Louis, Missouri
  - Cincinatti Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Background] Eghtesady P. Hypoplastic left heart syndrome: Rheumatic heart disease of the fetus? Med Hypotheses. 2006;66(3):554-65. doi: 10.1016/j.mehy.2005.09.013. Epub 2005 Oct 20. PMID 16242853
- [Background] McGregor KF, Spratt BG, Kalia A, Bennett A, Bilek N, Beall B, Bessen DE. Multilocus sequence typing of Streptococcus pyogenes representing most known emm types and distinctions among subpopulation genetic structures. J Bacteriol. 2004 Jul;186(13):4285-94. doi: 10.1128/JB.186.13.4285-4294.2004. PMID 15205431